CLINICAL TRIAL: NCT04519866
Title: A Randomized Controlled Trial of Electroacupuncture in the Management of Patients With Axial Spondyloarthritis in Singapore (E-AcuSpA)
Brief Title: Clinical Trial of Electroacupuncture in Axial Spondyloarthritis (E-AcuSpA)
Acronym: E-AcuSpA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); National University of Singapore (Other); Thong Chai Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/2435
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Spondylarthritis; Axial Spondyloarthritis
Keywords: Acupuncture; Electroacupuncture; Manual acupuncture
MeSH Terms: conditions — Spondylarthritis; Axial Spondyloarthritis | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): In addition to usual rheumatological care, patients in the electroacupuncture arm will undergo 2 courses of electroacupuncture treatment. Each treatment course will consist of 10 acupuncture sessions held over 5 weeks. Patient will take a break of 5-7 days in between each course of acupuncture.
  Interventions: Other: Electroacupuncture
- Manual acupuncture (Active Comparator): In addition to usual rheumatological care, patients in the manual acupuncture arm will undergo 2 courses of manual acupuncture treatment. Each treatment course will consist of 10 acupuncture sessions held over 5 weeks. Patient will take a break of 5-7 days in between each course of acupuncture.
  Interventions: Other: Manual acupuncture

INTERVENTIONS:
Other: Electroacupuncture — Manual acupuncture (see procedures below) will be administered first to obtain the "de qi" sensation. After "de qi" is obtained, the electroacupuncture unit will be connected to 1-3 pairs of acupoints. Current intensity used will be based on the tolerance of each patient. Needles with electrical stimulation will be retained for 30 min.
  Main acupoints will be Jingjin points (meridian sinews) along the Bladder meridian of Foot - Taiyang, such as Shenshuci, as well as Jingjin points (meridian sinews) at transverse process from L2 to L4, iliac crest and spinous process from S1 to S4. Secondary acupoints will also be selected based on patients' syndromes and symptoms.
  Arms: Electroacupuncture
Other: Manual acupuncture — After disinfecting the acupuncture points, acupuncture will be performed with the patient lying prone. Depending on the acupuncture points, 0.25mm X 25-75 mm sterile acupuncture needle will be used. Needles will be inserted 10-50 mm and either rotating manipulation or lifting-thrusting manipulation will be used to achieve "de qi" (a compositional sensation including soreness, numbness, distention and heaviness).
  Acupoints used will be similar to those mentioned for electroacupuncture (see above).
  Arms: Manual acupuncture

SUMMARY:
Axial spondyloarthritis (AxSpA) is a chronic disease that causes severe disability and poor quality of life. Current treatment options are limited and there are still significant non-responders to current western medications. Manual acupuncture has been shown to reduce pain in patients with AxSpA. There have been reports of electroacupuncture demonstrating more sustained pain relief. Therefore, the investigators aim to determine the clinical effectiveness, safety and cost-effectiveness of electroacupuncture as compared to manual acupuncture for patients with AxSpA through a randomized controlled trial.

DETAILED DESCRIPTION:
Patients with active axial spondyloarthritis despite non-steroidal anti-inflammatory drugs (NSAIDs) or biologics, will be randomly allocated to receive electroacupuncture or manual acupuncture on a 1:1 basis via random permuted block randomization. All patients will receive their standard of care (drug therapy and physiotherapy) as background therapy. This study will not be investigating any therapeutic or medicinal products (drugs).

Primary outcome would be the mean difference in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score between the 2 groups over 12 weeks (as assessed at weeks 0, 3, 6, 9, 12) adjusted for baseline covariate and other potential confounders. Patients will be followed up for BASDAI, other clinical, quality of life (QoL), economic outcomes as well as Traditional Chinese Medicine (TCM) syndrome scores over time for secondary and exploratory outcomes. A cost-effectiveness analysis will be performed. Adverse events will be recorded.

The primary hypothesis is that electroacupuncture may result in better disease activity control in patients with AxSpA as compared to manual acupuncture over 12 weeks, while secondary hypothesis is that electroacupuncture may result in greater improvements in other clinical and quality of life outcomes as compared to those receiving manual acupuncture over 24 weeks. The investigators also hypothesize that there is no difference in safety between both arms.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 years of age or older
* Diagnosed with AxSpA according to the 2009 Assessment of Spondyloarthritis International Society (ASAS) criteria
* Bath AS Disease Activity Index (BASDAI) score ≥4 on a 11-point Numerical Rating Scale (NRS)
* Failed 2 sequential NSAIDs (including cyclooxygenase-2 inhibitor) at maximal tolerated doses for ≥4 weeks in total
* Patients on concomitant biological therapy (e.g. tumour necrosis factor inhibitor therapy, anti-interleukin 17) or non-biologic disease-modifying antirheumatic drugs (DMARDs) (e.g. methotrexate (MTX) or sulfasalazine (SSZ) or leflunomide (LEF)) at study entry must be on the drug for ≥12 weeks and at stable dose for ≥4 weeks prior to randomisation
* Patients taking systemic corticosteroids have to be on stable dose of ≤10mg/day prednisolone or equivalent for at least two weeks before randomisation.

Exclusion Criteria:

* Pregnant or breastfeeding women
* With bleeding disorders
* With blood-borne communicable diseases (e.g. hepatitis B, hepatitis C, human immunodeficiency virus, etc)
* With implantable electrical device (e.g. pacemaker)
* Suffering from impaired skin sensation or serious skin lesions along the vertebrae

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mean difference in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score between both groups | Week 3, 6, 9, 12
  Mean difference in BASDAI score between both groups from baseline to weeks 3, 6, 9 and 12.
  BASDAI score ranges from 0-10, with higher scores indicating higher disease activity.

SECONDARY OUTCOMES:
Mean difference in Bath Ankylosing Spondylitis Functional Index (BASFI) score between both groups | Week 6, 12, 24
  Mean difference in BASFI score between both groups from baseline to weeks 6, 12 and 24.
  BASFI score ranges from 0-10, with higher scores indicating poorer functioning.
Mean difference in Bath Ankylosing Spondylitis Patient Global score (BAS-G) between both groups | Week 6, 12, 24
  Mean difference in BAS-G score between both groups from baseline to weeks 6, 12 and 24.
  BAS-G score ranges from 0-10, with higher scores reflecting poorer well-being.
Mean difference in Assessment of Spondyloarthritis International Society Health Index (ASAS HI) score between both groups | Week 6, 12, 24
  Mean difference in ASAS HI score between both groups from baseline to weeks 6, 12 and 24.
  ASAS HI score ranges from 0-17, with higher scores indicating poorer health status.
Mean difference in Ankylosing Spondylitis Quality of Life (ASQoL) score between both groups | Week 6, 12, 24
  Mean difference in ASQoL score between both groups from baseline to weeks 6, 12 and 24.
  ASQoL score ranges from 0-18, with higher scores indicating worse quality of life.
Mean difference in EuroQol- 5 Dimension (EQ-5D) score between both groups | Week 6, 12, 24
  Mean difference in EQ-5D score between both groups from baseline to weeks 6, 12 and 24.
  EQ-5D consists of a descriptive system and a visual analogue scale. The descriptive system covers 5 dimensions: mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression. Each dimension has a minimum and maximum score of 1 and 5 respectively, with higher scores representing a greater problem in that dimension. The visual analogue scale ranges from 0-100, with lower scores indicating poorer health status.
Mean difference in Work Productivity and Activity Impairment (WPAI) score between both groups | Week 6, 12, 24
  Mean difference in WPAI score between both groups from baseline to weeks 6, 12 and 24.
  WPAI measures absenteeism, presenteeism, work productivity loss and activity impairment. These are expressed as percentages, from 0-100, with higher numbers indicating greater impairment and less productivity.
Mean difference in healthcare costs between both groups | Week 6, 12, 24
  Mean difference in healthcare costs will be assessed for both groups at weeks 6, 12 and 24.
Mean difference in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score between both groups | Week 24
  Mean difference in BASDAI score between both groups from baseline to week 24. BASDAI score ranges from 0-10, with higher scores indicating higher disease activity.

OTHER OUTCOMES:
Mean difference in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score between both groups | Week 52
  Mean difference in BASDAI score between both groups from baseline to week 52. BASDAI score ranges from 0-10, with higher scores indicating higher disease activity.
Mean difference in Bath Ankylosing Spondylitis Functional Index (BASFI) score between both groups | Week 52
  Mean difference in BASFI score between both groups from baseline to week 52. BASFI score ranges from 0-10, with higher scores indicating poorer functioning.
Mean difference in Bath Ankylosing Spondylitis Patient Global score (BAS-G) between both groups | Week 52
  Mean difference in BAS-G score between both groups from baseline to week 52. BAS-G score ranges from 0-10, with higher scores reflecting poorer well-being.
Mean difference in Assessment of Spondyloarthritis International Society Health Index (ASAS HI) score between both groups | Week 52
  Mean difference in ASAS HI score between both groups from baseline to week 52. ASAS HI score ranges from 0-17, with higher scores indicating poorer health status.
Mean difference in Ankylosing Spondylitis Quality of Life (ASQoL) score between both groups | Week 52
  Mean difference in ASQoL score between both groups from baseline to week 52. ASQoL score ranges from 0-18, with higher scores indicating worse quality of life.
Mean difference in EuroQol- 5 Dimension (EQ-5D) score between both groups | Week 52
  Mean difference in EQ-5D score between both groups from baseline to week 52. EQ-5D consists of a descriptive system and a visual analogue scale. The descriptive system covers 5 dimensions: mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression. Each dimension has a minimum and maximum score of 1 and 5 respectively, with higher scores representing a greater problem for that dimension. The visual analogue scale ranges from 0-100, with lower scores indicating poorer health status.
Mean difference in Work Productivity and Activity Impairment (WPAI) score between both groups | Week 52
  Mean difference in WPAI score between both groups from baseline to week 52. WPAI measures absenteeism, presenteeism, work productivity loss and activity impairment. These are expressed as percentages, from 0-100, with higher numbers indicating greater impairment and less productivity.
Mean difference in healthcare costs will be assessed for both groups | Week 52
  Mean difference in healthcare costs will be assessed for both groups at week 52.
Mean difference in Traditional Chinese Medicine (TCM) syndrome scores will be assessed for both groups | Week 3, 6, 9, 12
  Mean difference in TCM syndrome scores will be assessed for both groups at weeks 0, 3, 6, 9, and 12.
  In this study, the main TCM syndromes are: 1) Yang" deficiency in kidneys and "Du" meridian, 2) Deficiency in liver and kidney, 3) Blockage due to stagnated blood, 4) Blockage due to damp heat syndrome, and 5) Blockage due to damp cold syndrome.
  Each symptom under the syndromes has a minimum score of 0 and maximum score of 3, with higher scores indicating greater symptom severity. Scores would be added up to tabulate syndrome scores, with higher scores indicating greater syndrome severity.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Fong, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwan YH, Fong W, Ang XL, Tan CS, Tai BC, Huang Y, Bilger M, Phang JK, Tan HC, Lee JV, Sun L, Tan CT, Dong BQ, Koh HL, Leung YY, Lui NL, Yeo SI, Ng SC, Fong KY, Thumboo J, Ostbye T. Traditional Chinese medicine (TCM) collaborative care for patients with axial spondyloarthritis (AcuSpA): protocol for a pragmatic randomized controlled trial. Trials. 2019 Jan 14;20(1):46. doi: 10.1186/s13063-018-3117-2. PMID 30642381

DOCUMENTS (2):
  • Study Protocol (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT04519866/Prot_002.pdf
  • Informed Consent Form (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT04519866/ICF_001.pdf